CLINICAL TRIAL: NCT01131624
Title: An Open-label, Multicentre, Randomised, 2-arm Study to Investigate the Comparative Efficacy and Safety of Intravenous Ferric Carboxymaltose Versus Oral Iron for the Treatment of Iron Deficiency Anaemia in Pregnant Women
Brief Title: Comparative Efficacy and Safety of Intravenous Ferric Carboxymaltose (FCM) Versus Oral Iron for Iron Deficiency Anaemia in Pregnant Women
Acronym: ASAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vifor Pharma (Industry)
Collaborators: Pierrel Research Europe GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FER-ASAP-2009-01
Record Dates: First submitted 2010-05-25; First posted 2010-05-27 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2014-12

CONDITIONS: Anaemia
Keywords: Iron deficiency
MeSH Terms: conditions — Anemia; Iron Deficiencies | interventions — ferrous sulfate; Iron; ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferric carboxymaltose (Active Comparator): Subjects with bw ≥66 kg will receive an infusion of 1,000 mg iron as FCM and after 1 week a further 500 mg iron as FCM, depending on Hb at screening.
  subjects with bw <66 kg, 2-3 infusions of 500 mg iron as FCM will be administered within 2 weeks from baseline, depending on Hb at screening
  Interventions: Drug: Ferinject
- Oral Iron (Active Comparator): Oral Iron oral iron preparation will be provided at 200 mg iron per day in a convenient dosage schedule.
  Interventions: Drug: ferrous sulphate

INTERVENTIONS:
Drug: ferrous sulphate — 200 mg iron per day in a convenient dosage schedule.
  Other Names: Oral Iron
  Arms: Oral Iron
Drug: Ferinject — 1000-1500mg diluted only in sterile 0.9% sodium chloride, The maximum single dose of FCM that can be administered by intravenous infusion is 20 mL (1,000 mg iron) but should not exceed 15 mg of iron per kg of body weight. This means that for subjects with a bw below 66 kg a maximal dose of 500 mg iron per infusion is allowed.
  Other Names: Ferric carboxymaltose; FCM
  Arms: Ferric carboxymaltose

SUMMARY:
The purpose of this study is to look at how well Ferric Carboxymaltose, an intravenous iron therapy (iron that is infused directly into your body through a vein), compares with ferrous sulphate capsules taken by mouth in the treatment of iron deficiency anaemia during pregnancy.

DETAILED DESCRIPTION:
This is an open-label, multicentre, randomised, 2-arm study to assess the efficacy and safety of FCM compared to oral iron in pregnant women with IDA.

During the screening period (Days -10 to 0 before randomisation), subjects will be selected based on eligibility criteria. Subjects who meet all of the inclusion criteria and none of the exclusion criteria will undergo baseline assessments at baseline (Day 0) prior to the first dose of study medication.

Subjects will be randomised to receive either intravenous (IV) iron (FCM, 1,000-1,500 mg) or oral iron (ferrous sulphate, 100 mg iron twice a day; total dose 200 mg/day).

The treatment period will begin with the infusion of FCM or the intake of oral iron on Day 0.

All subjects will return for assessment of efficacy and safety at Weeks 3, 6, 9, 12 and at delivery (or whichever comes first).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged ≥18, gestational week ≥20, ≤33 at baseline visit with normal antenatal screening test results.
* Iron deficiency anaemia defined as Hb concentration ≥8 g/dl and ≤10.4 g/dL and serum ferritin ≤20 mcg/L at screening.
* Demonstrated the ability to understand the requirements of the study, abide by the study restrictions, and agree to return for the required assessments. Patients (or their representative) must provide written informed consent for their participation in the study.

Exclusion Criteria:

* Blood transfusion, erythropoietin treatment, parenteral iron or oral iron treatment (1 month prior to screening) or anticipated need for a blood transfusion during the study.
* Anaemia not caused by iron deficiency (e.g., aplastic, megaloblastic or haemolytic anaemia) or related to acute or ongoing, haemoglobinopathies, rheumatic and other chronic diseases, autoimmune diseases, malignancies, bone marrow diseases, enzyme defects and drug induced anaemia.
* Acute or chronic infection, clinically relevant active inflammatory disease (C-reactive protein >10 mg/dl or outside reference range), any acute infection at screening.
* Pre-eclampsia.
* Multiple pregnancy.
* Evidence on any significant abnormalities on anomaly ultrasound.
* Haemochromatosis or other iron storage disorders.
* Folate deficiency (S-folate <4.5 nmol/L) at screening.
* Vitamin B12 deficiency (S-cobalamin <145 pmol/L) at screening.
* Serious medical condition, uncontrolled systemic disease or any other medical condition that, in the judgment of the Investigator, prohibits the patient from entering or potentially completing the study.
* Known chronic renal failure (defined as creatinine clearance <30 mL/min calculated by Cockcroft-Gault or modification of diet in renal disease formula).
* Severe cardiovascular diseases.
* Known human immunodeficiency virus/acquired immunodeficiency syndrome, hepatitis B virus or hepatitis C virus infection.
* Inability to fully comprehend and/or perform study procedures in the Investigator's opinion
* History of endocrine disorders
* Ongoing significant neurological or psychiatric disorders including psychotic disorders or dementia
* Recent significant bleeding/surgery (within the 3 months prior to screening).
* Chronic/acute hepatic disorder or elevating of liver enzymes (aspartate aminotransferase, alanine aminotransferase) over 2 times above the upper normal limit at screening.
* Participation in any other interventional study since estimated conception and throughout study participation.
* Known hypersensitivity to FCM or other IV iron preparations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2010-05; Primary Completion 2014-05 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Average Hb increase after 3 weeks in FCM compared to oral iron treated subjects (superiority). | 3 weeks after baseline

SECONDARY OUTCOMES:
Change in Hb from baseline at Week 6 | 6 weeks after baseline
Change in Hb from baseline at Week 9 | 9 weeks after baseline
Change in Hb from baseline at Week 12 | 12 weeks after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christian Breymann, Principal Investigator — University of Zurich
Locations (20):
- The Northern Hospital, Epping, Victoria, Australia
- Germany (3):
  - Vivantes Klinikum Neukölln, Klinikum für Geburtsmedizin, Berlin
  - Klinik Für Frauenheilkunde und Geburtshilfe Universitätsklinikum Marburg, Marburg
  - Perinatalzentrum, Klinikum Innenstadt LMU, München
- Sweden (5):
  - Kvinnokliniken, Falu lasarett, Falun
  - Kvinnokliniken, University Hospital, Lund
  - Kvinnokliniken, Karolinska University Hospital, Stockholm
  - Karolinska Universitetssjukhuset Huddinge, Centrum för fostermedicin KK, Stockholm
  - University Hospital, Dept of obstetrics and gynecology Uppsala, Uppsala
- Switzerland (7):
  - Universitätsspital Basel, Geburtshilfe und Schwangerschaftsmedizin Frauenklinik, Basel
  - Inselspital, Department of Obstetrics and Gynecology, Bern
  - Humboldtstrasse, Bern
  - HUG, Département de Gynécologie-Obstétrique, Geneva
  - CHUV, Département de Gynécologie-Obstétrique, Lausanne
  - OR Lugano, sede Ospedale Civico, Clinica ginecologia ostetricia, Lugano
  - Universitätsspital Zürich, Departement Frauenheilkunde, Zurich
- Turkey (Türkiye) (4):
  - Cukurova University Hospital, Adana
  - Istanbul Uni. Ist. Med. Faculty, Istanbul
  - Zeynep Kamil Hospital, Arakiyeci Haci Mehmet Mahallesi., Istanbul
  - Dr. Kutfi Kirdar Kartal Research and Education Hospital, Istanbul